CLINICAL TRIAL: NCT04782050
Title: Diagnostic échographique Non-invasif Des Maladies Chroniques du Foie en Consultation d'hépatologie
Brief Title: Non-invasive Ultrasound Diagnosis of Chronic Liver Diseases in Hepatology Consultation
Acronym: DIACEPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: E-Scopics (Industry)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ES201; 2021-A00612-39 (Other: ANSM (France - n°IDRCB)); 21.01563.000015 (Other: Ethical committee CPP Est I)
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Liver Diseases; Liver Cirrhosis; Non-Alcoholic Fatty Liver Disease
Keywords: Elastography; Attenuation; Sound speed; Ultrasound
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Intervention Model Description: All patients recruited will receive routine care for liver assessment followed by an exam using the device subject of the research.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental)
  Interventions: Device: Ultrasound liver assessment

INTERVENTIONS:
Device: Ultrasound liver assessment — The intervention consists in an ultrasound exam performed with the ultrasound medical device subject of the research.
  Other Names: Elastography; Ultrasound attenuation; Sound speed

SUMMARY:
Early screening and monitoring of chronic liver diseases in hepatology practice has become crucial. To achieve this goal, hepatology clinics need simple and available tools at the point-of-care to perform disease severity assessment. The objective of this study is to assess the performance of a new non-invasive ultrasound-based system for the assessment of liver fibrosis and steatosis severity, via ultrasound biomarkers such as tissue stiffness (correlated to fibrosis severity) and ultrasound tissue attenuation (correlated to steatosis extent).

DETAILED DESCRIPTION:
The study will enroll adult patients with known chronic liver disease, and referred to a hepatology outpatient visit for liver fibrosis assessment.

Performances will be assessed from correlation coefficients between biomarkers estimated by the medical device subject of the research and reference measurements obtained non-invasively from other commercially available equipment.

Repeatability and reproducibility of biomarkers estimations by the medical device subject of the research will be assessed from intraclass correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with known chronic liver disease and referred to the outpatient hepatology clinic for a consultation focused on chronic liver disease severity assessment, independently of the study (=in routine patient care).
* Patient who voluntarily consents to participate in the study, after being informed on study objectives and personal rights
* Patient who is registered to the French social security program

Exclusion Criteria:

* Adult patients under guardianship
* Adult patients not being under guardianship, unable to express consent for participation
* Pregnant women
* Breastfeeding women
* Patients under deprivation of liberty
* In-hospital patients not having given their consent to participate, or admitted in emergency
* Patients admitted in social and care centers for other reasons than those of the research
* Patients enrolled in other studies that have the potential to interfere with current research, or during the exclusion period forced by their participation in other research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Correlation of biomarkers to existing biomarker references | At study completion, 1 year
  Biomarkers measurements performed with the device subject of the research and commercially available equipment (2 other devices used in routine care) will be compared by analysis of correlation. The analysis outcome will be the R² coefficient and its p value.
Diagnostic performance of biomarkers in research | At study completion, 1 year
  Area under the receiver operating characteristic (ROC) curve will be used an a general assessment of diagnostic performance against dichotomized population according to commercially available diagnostic biomarkers.
  Conventional diagnostic estimators in the studied population will be derived from the ROC analysis: sensitivity, specificity, positive and negative predictive values, and diagnostic accuracy.

SECONDARY OUTCOMES:
Repeatability intraclass correlation coefficients (ICC) | At study completion, 1 year
  Repeatability will be assessed by calculating the ICC across 2 series of measurements performed by the same operator.
Reproducibility intraclass correlation coefficients (ICC) | At study completion, 1 year
  Reproducibility will be assessed by calculating the ICC across 2 series of measurements performed by 2 different operators.

CONTACTS AND LOCATIONS:
Overall Officials: Victor de Lédinghen, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France